CLINICAL TRIAL: NCT01972906
Title: Traditional Chinese Moxibustion for Primary Dysmenorrhea
Brief Title: Moxibustion for Primary Dysmenorrhea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011SZ0302
Record Dates: First submitted 2013-10-22; First posted 2013-10-31 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Primary Dysmenorrhea
Keywords: moxibustion; primary dysmenorrhea
MeSH Terms: interventions — Moxibustion; fenbid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxibustion treatment group (Experimental): Apply traditional acupuncture to prevent the dysmenorrhea according to traditional Chinese medicine theory
  Interventions: Device: moxibustion
- Medicine control group (Active Comparator): Ibuprofen Sustained Release Capsules will be penetrated for dysmenorrhea
  Interventions: Drug: Ibuprofen Sustained Release Capsules

INTERVENTIONS:
Device: moxibustion — apply moxibustion according to traditional Chinese medicine
  Arms: Moxibustion treatment group
Drug: Ibuprofen Sustained Release Capsules — apply Ibuprofen (H20013062), 0.3g， Bid, lasting 3 days before menstrual cycle
  Other Names: Fenbid
  Arms: Medicine control group

SUMMARY:
Hypothesis: Moxibustion is effective for managing primary dysmenorrhea. Aim: To attest the effectiveness and safety of moxibustion for primary dysmenorrhea. Design: A randomized controlled trial. 152 participants will be included. Two arms: moxibustion treatment group and ibuprofen control group.

DETAILED DESCRIPTION:
There is no convincing evidence for the efficacy of moxibustion for primary dysmenorrhea, due to low methodologic quality and small sample size. The investigators designed the random clinical trial to investigates the effectiveness of moxibustion in treating primary dysmenorrhea, the purpose of this study is to provide the research base of moxibustion efficacy. The investigators also examined the acceptability and any adverse effects associated with the use of moxibustion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Guidelines of Primary dysmenorrhea clinical by the Society of Obstetricians and Gynaecologists of Canada
* Menstrual cycle is regular (28±7) days
* Syndrome differentiation of Traditional Chinese Medicine: Congealing cold-damp and Qi-stagnation and blood stasis
* Mean value of ≥40mm during last 3 months
* Informed consent form must be signed by patient or lineal relative

Exclusion Criteria:

* Patients with secondary dysmenorrhea, which is caused by endometriosis, pelvic inflammation, myoma of uterus and so on
* Patients who are unconscious and psychotic
* Patients with serious primary illness or diseases of cardiovascular, liver, renal, gastrointestinal, hematological systems and so on
* Patients take prostaglandin synthetase inhibitors (PGSI) 2 weeks before inclusion
* Pregnant women or women in lactation

Ages: 13 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in menstrual pain intensity measured by VAS at 6 months | at baseline, 1st, 2nd, 3rd, 4th, 5th, 6th menstrual cycle after inclusion
  to assess the degree of dysmenorrhea

SECONDARY OUTCOMES:
Laboratory index-1 | at baseline, 4th menstrual cycle after inclusion
  prostaglandin (PGF2a、PGE2)
Cox Menstrual Symptom Scale Cox Menstrual Symptom Scale | 1st, 2nd, 3rd, 4th, 5th, 6th, 7th menstrual cycle after inclusion
  to assess the change of symptom during menstrual cycle
Laboratory Index-2 | at baseline, 4 menstrual cycles after inclusion
  oxytocin
Laboratory Index-3 | at baseline, 4 menstrual cycles after inclusion
  β-endorphin
Laboratory Index-4 | at baseline, 4 menstrual cycles after inclucion
  plasma endothelin-1
Laboratory Index-5 | at baseline, 4 menstrual cycles after inclusion
  nitric oxide
Laboratory Index-6 | at baseline, 4 menstrual cycles after inclusion
  Plasma vascular pseudohemophilia factors

CONTACTS AND LOCATIONS:
Overall Officials: Fanrong Liang, Professor, Principal Investigator — Chengdu University of TCM
Locations (1):
- Affiliated hospital of Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Yang M, Chen X, Bo L, Lao L, Chen J, Yu S, Yu Z, Tang H, Yi L, Wu X, Yang J, Liang F. Moxibustion for pain relief in patients with primary dysmenorrhea: A randomized controlled trial. PLoS One. 2017 Feb 7;12(2):e0170952. doi: 10.1371/journal.pone.0170952. eCollection 2017. PMID 28170396